CLINICAL TRIAL: NCT05027763
Title: Can Low-fat/high-fiber or Fermented Diet Modulate the Gut Microbiome to Improve Surgical Outcomes?
Brief Title: Effect of Preoperative Diet on Perioperative Gut Microbiome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cindy Kin, Assistant Professor of Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 62330
Record Dates: First submitted 2021-08-17; First posted 2021-08-30 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-03

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Arm (No Intervention): Standard care - patients will not receive specific dietary advice.
- High Fiber/low fat (Experimental): Patients will receive sample meals and education/support, will be asked to follow this diet for 10 days.
  Interventions: Behavioral: high-fiber/low fat
- Fermented (Experimental): Patients will receive sample meals and education/support, will be asked to follow this diet for 10 days.
  Interventions: Behavioral: fermented

INTERVENTIONS:
Behavioral: high-fiber/low fat — high fiber/low fat preoperative diet
  Arms: High Fiber/low fat
Behavioral: fermented — fermented preoperative diet
  Arms: Fermented

SUMMARY:
The aim of the study is to evaluate the gut microbiome (i.e. bacteria, viruses, and fungi that reside in the gut) of people undergoing abdominal surgery, evaluate whether specific diets can change the gut microbiome, and, if so, whether those changes translate into better surgical outcomes.

DETAILED DESCRIPTION:
Standard of care: patients undergoing major abdominal colorectal surgery are sometimes advised to eat healthfully prior to surgery, but without more specific recommendations regarding their diet.

Research Activities:

1. Screening: eligible patients will be identified through screening the clinic schedules.
2. Enrollment: in person or remotely, after the patient is determined to require major abdominal surgery, they will be invited to participate in the study. If they consent to participate, they will be randomized to receive either low-fat/high-fiber diet, high-fermented diet, or continue with their normal diet for 10-14 days prior to the surgery.
3. Intervention: at baseline, data will be collected regarding clinical information of the patients (age, body mass index, comorbidities, medications or supplements, physical activity levels, antibiotic or probiotic use in the past six months), and baseline dietary pattern, which will be evaluated through application of a validated Food Frequency Questionnaire (DHQ III). Patients in the intervention arms (low- fat/high-fiber diet or high-fermented diet) will receive meal samples during the 10-14 days preceding surgery. Patients in the control arm will receive a $25 grocery voucher. Adherence to the diet will be assessed through regular check ins with the patients.

   Stool samples will be collected in five timepoints: at the beginning of the study, after the dietary intervention, during surgery, in the first week after the surgery, and between 21-30 days after surgery. The stool samples will be sent for analysis of the microbiome.

   A fragment of the resected bowel will also be sent for analysis of the mucosal-associated microbiome.
4. Closeout: After surgery, all patients will receive the same standard dietary protocol and care, and will be followed for 30 days without any further intervention.

ELIGIBILITY:
Inclusion Criteria:

* undergoing major abdominal colorectal surgery with intestinal resection in 2 or more weeks

Exclusion Criteria:

* patients who do not speak English or Spanish
* houseless patients
* decisionally impaired patients
* presence of ileostomy prior to the surgical procedure
* surgery without intestinal resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiome alpha and beta diversity according to pre-operative diet intervention | Two weeks prior to surgery
  Metagenomic sequencing will be performed on stool samples before and after dietary change.

SECONDARY OUTCOMES:
Change in gut microbiome alpha and beta diversity after surgery according to pre-operative diet | Surgery date until 1 month after surgery
  Metagenomic sequencing will be performed on stool samples collected in the first week after surgery and 30 days after surgery
Frequency and severity of surgical complications according to pre-operative diet | 30 days after surgery
  Comprehensive Complication Index (CCI) score will be used to measure number and severity of surgical complications occurring within 30 days after surgery. Comprehensive Complication Index score includes minimum value of 0 and maximum value of 100; higher score means higher severity of complication(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyoju SK, Adriaansens C, Wienholts K, Sharma A, Keskey R, Arnold W, van Dalen D, Gottel N, Hyman N, Zaborin A, Gilbert J, van Goor H, Zaborina O, Alverdy JC. Low-fat/high-fibre diet prehabilitation improves anastomotic healing via the microbiome: an experimental model. Br J Surg. 2020 May;107(6):743-755. doi: 10.1002/bjs.11388. Epub 2019 Dec 26. PMID 31879948
- [Background] Kok DE, Arron MNN, Huibregtse T, Kruyt FM, Bac DJ, van Halteren HK, Kouwenhoven EA, Wesselink E, Winkels RM, van Zutphen M, van Duijnhoven FJB, de Wilt JHW, Kampman E. Association of Habitual Preoperative Dietary Fiber Intake With Complications After Colorectal Cancer Surgery. JAMA Surg. 2021 Jun 16;156(9):1-10. doi: 10.1001/jamasurg.2021.2311. Online ahead of print. PMID 34132738
- [Background] Wastyk HC, Fragiadakis GK, Perelman D, Dahan D, Merrill BD, Yu FB, Topf M, Gonzalez CG, Van Treuren W, Han S, Robinson JL, Elias JE, Sonnenburg ED, Gardner CD, Sonnenburg JL. Gut-microbiota-targeted diets modulate human immune status. Cell. 2021 Aug 5;184(16):4137-4153.e14. doi: 10.1016/j.cell.2021.06.019. Epub 2021 Jul 12. PMID 34256014
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846